CLINICAL TRIAL: NCT07066865
Title: Safety and Efficacy of Sutureless Dehydrated Amniotic Membrane (Omnigen) Mounted on Contact Lens (Omnilenz) for Ttt of Ocular Graft vs Host Disease
Brief Title: Evaluation of the Safety and Effectiveness of omniLenz in Patient With Ocular Graft vs Host Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Farwaniya Hospital (Other Government)
Responsible Party: Principal Investigator, Nancy Lotfy, MD, MD, Farwaniya Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1630/2025
Record Dates: First submitted 2025-06-19; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-06

CONDITIONS: Ocular Graft Versus Host Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patient who applied OmniLenz for one week (Experimental)
  Interventions: Device: omniLenz

INTERVENTIONS:
Device: omniLenz — sutureless dehydrated amniotic membrane (omnigen) mounted on contact lens (omnilenz)

SUMMARY:
A case series of patients presented with graft versus host disease with ocular involvement . The study recruited a total of 3 patients who were referred to cornea clinic of Farwaniya Hospital, Kuwait between April 2022 and April 2024. All cases presented with severe dryness, spks and corneal epithelial defect not responding to other measures of treatment. An OmniLenz was applied for each patient for one week. Primary outcome measures included healing of the corneal resistant epithelial defect, secondary outcome measures were improvement of signs of dryness.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Ocular graft versus host disease

Exclusion Criteria:

- Patient with conjunctival fibrosis and symblephara formation (which interfere with application of the omnilenz)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Epithelial healing, Slit lamp examination with cobalt blue light after installation of fluorescein eye drops | 1 week ( duration of the application of omnilenz )

SECONDARY OUTCOMES:
Omnigen tolerability, Questionnaire for the patients asking about discomfort sensation or the need to patch the eye | 1 week ( duration of the application of omnilenz )

CONTACTS AND LOCATIONS:
Locations (1):
- Farwanyia Hospital, Al Farwānīyah, Kuwait